CLINICAL TRIAL: NCT05203848
Title: Community Dance Program (CDP) for Older Adults - a Pilot Randomized Control Trial
Brief Title: Community Dance Program (CDP) for Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Singapore (Other)
Collaborators: Lions Befrienders (Unknown)
Responsible Party: Principal Investigator, Vivien Xi WU, PhD, Assistant Professor, National University of Singapore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: NUS-IRB-2020-808
Record Dates: First submitted 2021-12-13; First posted 2022-01-24 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2022-01

CONDITIONS: Healthy Aging
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dance program intervention (Experimental): The community dance program (CDP) will be developed to promote older adults' physical and mental well-being through dancing. The contents of the program are developed based on the literature review (Rossberg-Gempton & Poole, 2008). The CDP will be delivered over a period of 8 weeks.
  Interventions: Procedure: Community Dance Intervention
- Control group (Placebo Comparator): There will be no dance intervention among control group participants.
  Interventions: Other: Control group

INTERVENTIONS:
Procedure: Community Dance Intervention — The main dance instructor for the CDP is Yarra Ileto, who is the Artistic Director for NUS Dance Synergy. Yarra was trained at LASALLE College of the Arts, graduating with a First Class BA (Hons) Dance in 2008. Also, she has experience with crafting and conducting Community Dance Programs (CDP) for Seniors. Yarra will be developing the dance lesson plan and also training selected students from NUS Dance Synergy to guide the seniors during the dance sessions. Older adults will learn and practice the basic steps together for the first few weeks. Then, the student dance instructors will start teaching the dance formation. During each session, participants will need to warm up first to prevent injuries before practicing dance steps. Small group practicing is reserved for older adults to interact with each other. All the participants will do relaxation exercises before ending the session to cool down their bodies and release muscle tensions.
  Arms: Dance program intervention
Other: Control group — Control group
  Arms: Control group

SUMMARY:
Objectives:

The primary objective of the proposed project is to develop and evaluate a Community Dance Program (CDP) for community-dwelling older adults, which is aimed at promoting physical strength, balance, cognition, mental and psycho-social well-being of the older adults. A distinctive feature of our project is that a team of researchers across disciplines and community partners will collaborate to develop the program and bring benefits to the older adults living in the community.

DETAILED DESCRIPTION:
Research Design:

The research design consists of: (1) Development and implementation of CDP. A pilot cluster randomized controlled trial (RCT) will be conducted to assess the feasibility and primary effect of the program in enhancing the physical, mental, cognitive, and psycho-social health, quality of life, and social support among older adults. (2) Process Evaluation, follow-up focus group discussions will be conducted to assess the acceptability, strengths and limitations of CDP based on the participants' perspectives.

Data Collection and Analysis:

A set of questionnaires will be administered to the older adults. The data will be collected at two time points: baseline and 8-week follow-up. Descriptive statistics, Paired sample t-test, Analysis of Covariance (ANCOVA), General Linear Model (GLM) will be used to examine the difference between the baseline and post-intervention to compare outcome measures from pre to post-implementation. The audio-recorded focused group discussion will be transcribed verbatim respectively. Thematic analysis will be applied to provide an in-depth and rich analysis of the verbatim.

Potential Impact:

CDP will make a positive impact on the older adults' physical, mental and psychological wellbeing. Those impacts will then encourage older adults to live an active life and maximize their social capital within the community. Therefore, CDP promotes the health and wellbeing of the community-dwelling older adults and reduces geriatric-related conditions. The outcome of the study will have tremendous potential to be implemented at a larger scale in the community. Upon completion of the project, the investigators will work closely with community centres and senior activity centres to integrate CDP into their existing programs. CDP could then benefit a larger population given the evidence gathered from this research to enhance the physical, mental and psychological wellbeing of the older adults.

ELIGIBILITY:
Inclusion Criteria:

* Aged 55 to 85
* Able to understand and communicate in either English or Mandarin
* Able to give consent to participate (have sufficient mental capacity as assessed by the MoCA, with a score of 16 and above)
* Lives within the community setting
* Able to ambulate with minimal assistance
* Able to commit a total of 8 hours over the 8-week period dancing program

Exclusion Criteria:

* Medical conditions which result in limitation of dancing
* Older adults with compromised balance and mobility (those who obtained a score of < 5 on the Short Physical Performance Battery (SPPB)
* Severe cognitive or psychiatric disorders
* Severe hearing or vision impairments
* Older adults from the control group who also participate in any other dance group during the intervention period
* Older adults who are uncomfortable with video-recording of the dance sessions

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2021-09-09 (Actual); Primary Completion 2022-12-21 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Physical health: Blood pressure | 3 months
  Blood pressure readings will be measured in units of millimeters of mercury (mmHg). Both systolic and diastolic blood pressure values will be recorded before versus after the research intervention to investigate for any significant changes.
Physical health: Body Mass Index (BMI) | 3 months
  BMI was obtained from each participant by measuring his/her height in units of meters and weight in units of kilograms, followed by this formula: kg/m^2. BMI values will be recorded before versus after the research intervention to investigate for any significant changes.
Physical health: Waist and hip circumferences | 3 months
  Waist and hip circumferences of each participant will be obtained in units of centimeters (cm). These values will be recorded before versus after the research intervention to investigate for any significant changes.
Physical health: Short Physical Performance Battery (SPPB) | 3 months
  SPPB is a comprehensive instrument that can be used to measure balance, mobility, and muscle strength in older adults. It consists of balance tests (i.e., side-by-side stand, semi-tandem stand, tandem stand), gait speed tests, and chair stand tests. All values will be recorded in units of seconds and consolidated into the corresponding sum of scores upon successful completion of each test. Higher SPPB scores indicate greater physical capabilities.
Psychosocial health: Subjective Happiness Scale | 3 months
  Subjective Happiness Scale using a "subjectivist" approach to the assessment of happiness, a 4-item measure of global subjective happiness was developed and validated in 14 studies with a total of 2732 participants (Lyubomirsky & Lepper,1999). A 7-point Likert scale (1 = less happy to 7 = more happy) was used, with higher scores indicating higher subjective happiness.
Cognitive health: Montreal Cognitive Assessment (MoCA) | 3 months
  MoCA was designed as a screening instrument for mild cognitive dysfunction. It assesses various cognitive domains including attention, concentration, executive function, memory, language, visuospatial, and arithmetic skills. The total possible score is 30 points, with the cutoff score of this research study being 16 points. Participants who scored below 16 points will not be included in the research study. A lower MoCA score indicates greater cognitive dysfunction.
Cognitive health: Symbol Digit Modalities Test (SDMT) | 3 months
  SDMT is a screening measure for cerebral dysfunction in adults. A coding key is presented consisting of nine abstract symbols, each paired with a number. The participant is required to scan through the coding key and write down the number corresponding to each symbol, as rapidly as possible. The number of correct answers within the 90-second interval is recorded. The maximum score is 110, with lower scores suggesting cerebral dysfunction.
Cognitive health: The Washington University Dementia Screening Test (AD8) | 3 months
  This scale is also known as "Eight-item Interview to Differentiate Aging and Dementia". The participant was asked to rate changes in his/her ability for each of the items, without attributing causability. The final score is computed by consolidating the sum of the items marked with a change due to cognitive problems, with higher scores indicating higher impairment in cognition.
Quality of Life: WHOQOL-AGE | 3 months
  WHOQOL-AGE is a self-reported questionnaire that was designed specifically to measure quality of life (QoL) in the older adult population (Caballero et al., 2013). It consists of 13 items which are selected from the other versions of WHOQOL instruments (5 items from WHOQOL-OLD and 8 items from EUROHIS-QOL). The items were assessed on a five-point Likert scale, ranging from 1 (very dissatisfied) to 5 (very satisfied), with higher scores suggesting higher QoL. WHOQOL-AGE has been evaluated and has shown good reliability and validity (Santos et al., 2018).
Physical health: DNA Methylation (DNAm) Testing | 3 months
  DNA Methylation (DNAm) Testing was conducted by collecting the participants' saliva into a 5 mL polypropylene tube. The participants were instructed to let saliva collect in their mouth and gently push the saliva into a short section of common drinking straw into the tube. Saliva samples were aliquoted into 2 mL polypropylene cryovials, with colour coded lids. De-identified samples will be stored at -80 degrees C. De-identified saliva samples were sent to Muhdo Health Pte Ltd, a UK-based epigenetics testing company for DNA extraction and whole epigenome sequencing, in which the results were shared to the research team.
Physical health: MOXY Near-Infrared Spectroscopy (NIRS) Measurement of muscle oxygenation | 3 months
  MOXY Near-Infrared Spectroscopy (NIRS) Measurement of muscle oxygenation was conducted by attaching a near-infrared spectroscopy probe (Moxy Monitor) on the belly of the vastus lateralis (quadriceps) muscle, midway between the lateral epicondyle and greater trochanter of the femur (DeLorey et al., 2004). This was performed to measure relative muscle oxygenation level before, during contraction, and for up to 1 hour post-exercise. The device measured muscle O2 saturation (SmO2) every 2 seconds throughout the trial, and has been validated and described in detail in a study by Crum et al. (2017). For the present study, the probe was placed on the participant's quadriceps muscle during the SPPB.

SECONDARY OUTCOMES:
Intergenerational communication | 3 months
  Global Perceptions of Intergenerational Communication Scale (GPIC) was developed by McCann & Giles (2007) to measure perceptions of intergenerational communicative experiences. It consists of 25 items rated on a 5-point scale (1 = strongly disagree; 5 = strongly agree). The first 14 items of the scale assess perceptions of others' communication while the remaining 11 items assess perceptions of one's own communication.
Social support | 3 months
  Social Support Questionnaire 6 items (SSQ6) was developed by Sarason and colleagues (Sarason, Sarason, Shearin & Pierce,1987). It is used to measure the number of person providing support to an individual and the satisfaction level of the individual who received the support. The scale consists of 6 items. Rating of the items is from 1 (very dissatisfied) to 6 (very satisfied). With excellent Cronbach alphas of 0.90 and 0.93 for 2 respective domains, the scale has been proved to be valid and reliable.
Sociodemographic data | 3 months
  Social-demographic data including age, gender, ethnicity, religion, marital status, employment status, education, social-economic status, source of financial support, household type/ownership, living arrangement and number of children will be collected.

CONTACTS AND LOCATIONS:
Locations (1):
- National University of Singapore, Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wu XV, Tam WSW, Yap XY, Zhang J, Mok WYJ, Lim ZX, Goh J. Intergenerational approach of community dance program for older adults in singapore: a feasibility cluster-controlled trial. BMC Geriatr. 2025 Dec 2;26(1):17. doi: 10.1186/s12877-025-06796-7. PMID 41327006